CLINICAL TRIAL: NCT02676180
Title: A Prospective Observational Study to Determine the Negative Predictive Value of UroMark to Rule Out the Presence of Bladder Cancer in Patients With Haematuria.
Brief Title: Detecting Bladder Cancer Using the UroMark Test.
Acronym: DETECT I
Status: Completed | Type: Observational
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 15/0883
Record Dates: First submitted 2015-12-18; First posted 2016-02-08 (Estimated); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Population Groups; Watchful Waiting

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples With DNA — Urine will be collected for analysis using UroMark assay.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Group
  Other Names: Observational

SUMMARY:
DETECT I is a prospective multicentre observational diagnostic study to assess the performance of the UroMark assay to rule out bladder cancer in patients with haematuria. The study will recruit consecutive patients attending haematuria clinics as well as patients referred to urology outpatient clinics for investigation of haematuria. Consenting patients will be provided with a urine sample collection kit and asked to provide a urine sample. An additional urine sample for control assay testing will be provided after the clinic attendance.

DETAILED DESCRIPTION:
Transitional cell carcinoma (TCC) of the urinary bladder is responsible for >12,000 new cases of cancer and >5,000 deaths per year in England and Wales. Most bladder cancers are non-muscle invasive bladder cancer (NMIBC) and do not invade deeply at presentation, but 80% of tumours recur within 3 years. For muscle invasive bladder cancer (MIBC), the 5 year survival is around 50%. Cystoscopy is the standard test for detection of bladder cancer along with imaging to assess the upper tracts and the common presenting symptom is haematuria. Cystoscopy is an invasive procedure and results in urinary infection in up to 5% of cases. Cystoscopy is performed under local anaesthetic and patients are required to attend hospital clinics for the test. About one in 10 patients who are investigated for haematuria will be found to have bladder cancer. Frequently, patients are not referred for investigation of haematuria at the time of first presentation and there is a delay in diagnosis of the disease. The early detection of bladder cancer by means of a non-invasive tumour marker test would impact on the management of the disease. There is an unmet need for a simple, non-invasive, highly sensitive and specific method for detecting bladder cancer.

This study will determine the accuracy of UroMark a high-throughput multiplex PCR test to detect bladder cancer in DNA from urine. The study will address the unmet clinical need to improve detection of bladder cancer. The rationale for the trial is based on proof of concept studies which provide compelling evidence that a panel of methylation markers can be applied to detect bladder cancer with high sensitivity and specificity. It will be also be possible to collect and store fractions of urine for assessment of other DNA related biomarkers as well as non-DNA assays for example cellular proteins, soluble biomarkers in urine supernatant and RNA transcripts in sediment cells. In this study we will compare the UroMark assay with established assays including urinary cytology, FISH as well as developing assays such as MCM5. In this proposal excess urine will be stored for these studies.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be over 18 years of age.
* Participants undergoing investigation for visible and non-visible haematuria.
* Able to give informed written consent.

Exclusion Criteria:

* Unwilling to have standard haematuria investigations.
* Unable to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with visible and non-visible haematuria (blood in urine) will be enrolled. About 10% of cases with haematuria will be found to have bladder cancer. For the majority of cases (60.5%), no cause is found. Other causes include stone disease (3.6%), benign prostate conditions (20-30%), renal disease (9.8%) infection (13%) and renal/prostate cancer (1%). The DETECT I study will determine if the UroMark test can be used to rule out bladder cancer in cases referred for investigation of haematuria.
Sampling Method: Non-Probability Sample
Enrollment: 3700 (Actual)
Dates: Start 2016-03-30 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Negative predictive value (NPV) of the UroMark test. | Baseline

SECONDARY OUTCOMES:
Negative predictive value (NPV) of control assay (FDA approved urinary marker (UroVision)). | Baseline
Negative predictive value (NPV) against imaging (ultrasound/CT) | Baseline
Negative predictive value (NPV) against combination of UroMark and imaging. | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: John Kelly, FRCS (urol), Principal Investigator — UCL
Locations (2):
- United Kingdom (2):
  - UCLH, London
  - James Cook University Hospital, Middlesbrough

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chan AW, Tetzlaff JM, Altman DG, Laupacis A, Gotzsche PC, Krleza-Jeric K, Hrobjartsson A, Mann H, Dickersin K, Berlin JA, Dore CJ, Parulekar WR, Summerskill WS, Groves T, Schulz KF, Sox HC, Rockhold FW, Rennie D, Moher D. SPIRIT 2013 statement: defining standard protocol items for clinical trials. Ann Intern Med. 2013 Feb 5;158(3):200-7. doi: 10.7326/0003-4819-158-3-201302050-00583. PMID 23295957
- [Background] Chan AW, Tetzlaff JM, Gotzsche PC, Altman DG, Mann H, Berlin JA, Dickersin K, Hrobjartsson A, Schulz KF, Parulekar WR, Krleza-Jeric K, Laupacis A, Moher D. SPIRIT 2013 explanation and elaboration: guidance for protocols of clinical trials. BMJ. 2013 Jan 8;346:e7586. doi: 10.1136/bmj.e7586. PMID 23303884
- [Background] Malmstrom PU, Sylvester RJ, Crawford DE, Friedrich M, Krege S, Rintala E, Solsona E, Di Stasi SM, Witjes JA. An individual patient data meta-analysis of the long-term outcome of randomised studies comparing intravesical mitomycin C versus bacillus Calmette-Guerin for non-muscle-invasive bladder cancer. Eur Urol. 2009 Aug;56(2):247-56. doi: 10.1016/j.eururo.2009.04.038. Epub 2009 Apr 24. PMID 19409692
- [Background] Lyratzopoulos G, Abel GA, McPhail S, Neal RD, Rubin GP. Gender inequalities in the promptness of diagnosis of bladder and renal cancer after symptomatic presentation: evidence from secondary analysis of an English primary care audit survey. BMJ Open. 2013 Jun 24;3(6):e002861. doi: 10.1136/bmjopen-2013-002861. PMID 23798742
- [Background] Mitra AP, Cote RJ. Molecular screening for bladder cancer: progress and potential. Nat Rev Urol. 2010 Jan;7(1):11-20. doi: 10.1038/nrurol.2009.236. PMID 20062071
- [Background] Sangar VK, Ragavan N, Matanhelia SS, Watson MW, Blades RA. The economic consequences of prostate and bladder cancer in the UK. BJU Int. 2005 Jan;95(1):59-63. doi: 10.1111/j.1464-410X.2005.05249.x. PMID 15638895
- [Background] Rodgers M, Nixon J, Hempel S, Aho T, Kelly J, Neal D, Duffy S, Ritchie G, Kleijnen J, Westwood M. Diagnostic tests and algorithms used in the investigation of haematuria: systematic reviews and economic evaluation. Health Technol Assess. 2006 Jun;10(18):iii-iv, xi-259. doi: 10.3310/hta10180. PMID 16729917
- [Background] Kelly JD, Fawcett DP, Goldberg LC. Assessment and management of non-visible haematuria in primary care. BMJ. 2009 Jan 16;338:a3021. doi: 10.1136/bmj.a3021. No abstract available. PMID 19151065
- [Background] Mowatt G, N'Dow J, Vale L, Nabi G, Boachie C, Cook JA, Fraser C, Griffiths TR; Aberdeen Technology Assessment Review (TAR) Group. Photodynamic diagnosis of bladder cancer compared with white light cystoscopy: Systematic review and meta-analysis. Int J Technol Assess Health Care. 2011 Jan;27(1):3-10. doi: 10.1017/S0266462310001364. Epub 2011 Jan 25. PMID 21262078
- [Background] Khadra MH, Pickard RS, Charlton M, Powell PH, Neal DE. A prospective analysis of 1,930 patients with hematuria to evaluate current diagnostic practice. J Urol. 2000 Feb;163(2):524-7. PMID 10647670
- [Background] Edwards TJ, Dickinson AJ, Natale S, Gosling J, McGrath JS. A prospective analysis of the diagnostic yield resulting from the attendance of 4020 patients at a protocol-driven haematuria clinic. BJU Int. 2006 Feb;97(2):301-5; discussion 305. doi: 10.1111/j.1464-410X.2006.05976.x. PMID 16430634
- [Background] Lotan Y, Elias K, Svatek RS, Bagrodia A, Nuss G, Moran B, Sagalowsky AI. Bladder cancer screening in a high risk asymptomatic population using a point of care urine based protein tumor marker. J Urol. 2009 Jul;182(1):52-7; discussion 58. doi: 10.1016/j.juro.2009.02.142. Epub 2009 May 17. PMID 19450825
- [Background] Hoque MO, Begum S, Topaloglu O, Chatterjee A, Rosenbaum E, Van Criekinge W, Westra WH, Schoenberg M, Zahurak M, Goodman SN, Sidransky D. Quantitation of promoter methylation of multiple genes in urine DNA and bladder cancer detection. J Natl Cancer Inst. 2006 Jul 19;98(14):996-1004. doi: 10.1093/jnci/djj265. PMID 16849682
- [Background] Dudderidge TJ, Kelly JD, Wollenschlaeger A, Okoturo O, Prevost T, Robson W, Leung HY, Williams GH, Stoeber K. Diagnosis of prostate cancer by detection of minichromosome maintenance 5 protein in urine sediments. Br J Cancer. 2010 Aug 24;103(5):701-7. doi: 10.1038/sj.bjc.6605785. Epub 2010 Jul 20. PMID 20648010
- [Background] Coenen MJ, Ploeg M, Schijvenaars MM, Cornel EB, Karthaus HF, Scheffer H, Witjes JA, Franke B, Kiemeney LA. Allelic imbalance analysis using a single-nucleotide polymorphism microarray for the detection of bladder cancer recurrence. Clin Cancer Res. 2008 Dec 15;14(24):8198-204. doi: 10.1158/1078-0432.CCR-08-1103. PMID 19088036
- [Derived] Tan WS, Ahmad A, Zhou Y, Nathan A, Ogunbo A, Gbolahan O, Kallam N, Smith R, Khalifeh M, Tan WP, Cohen D, Volanis D, Walter FM, Sasieni P, Kamat AM, Kelly JD. Hematuria Cancer Risk Score with Ultrasound Informs Cystoscopy Use in Patients with Hematuria. Eur Urol Oncol. 2025 Feb;8(1):87-93. doi: 10.1016/j.euo.2024.05.005. Epub 2024 May 28. PMID 38811250
- [Derived] Tan WS, Ahmad A, Feber A, Mostafid H, Cresswell J, Fankhauser CD, Waisbrod S, Hermanns T, Sasieni P, Kelly JD; DETECT I trial collaborators. Development and validation of a haematuria cancer risk score to identify patients at risk of harbouring cancer. J Intern Med. 2019 Apr;285(4):436-445. doi: 10.1111/joim.12868. Epub 2019 Jan 4. PMID 30521125
- [Derived] Tan WS, Sarpong R, Khetrapal P, Rodney S, Mostafid H, Cresswell J, Watson D, Rane A, Hicks J, Hellawell G, Davies M, Srirangam SJ, Dawson L, Payne D, Williams N, Brew-Graves C, Feber A, Kelly JD; DETECT I trial collaborators. Does urinary cytology have a role in haematuria investigations? BJU Int. 2019 Jan;123(1):74-81. doi: 10.1111/bju.14459. Epub 2018 Aug 29. PMID 30003675
- [Derived] Tan WS, Feber A, Sarpong R, Khetrapal P, Rodney S, Jalil R, Mostafid H, Cresswell J, Hicks J, Rane A, Henderson A, Watson D, Cherian J, Williams N, Brew-Graves C, Kelly JD; DETECT I trial collaborators. Who Should Be Investigated for Haematuria? Results of a Contemporary Prospective Observational Study of 3556 Patients. Eur Urol. 2018 Jul;74(1):10-14. doi: 10.1016/j.eururo.2018.03.008. Epub 2018 Apr 10. PMID 29653885
- [Derived] Tan WS, Feber A, Dong L, Sarpong R, Rezaee S, Rodney S, Khetrapal P, de Winter P, Ocampo F, Jalil R, Williams NR, Brew-Graves C, Kelly JD. DETECT I & DETECT II: a study protocol for a prospective multicentre observational study to validate the UroMark assay for the detection of bladder cancer from urinary cells. BMC Cancer. 2017 Nov 15;17(1):767. doi: 10.1186/s12885-017-3758-7. PMID 29141603